CLINICAL TRIAL: NCT02694861
Title: A Multi-Center Single Arm One Year Prospective Follow-Up of Patients Treated With the CryoLife CardioGenesis Holmium:YAG Laser System for Transmyocardial Revascularization (The TMR 365 Study)
Brief Title: CardioGenesis Transmyocardial Revascularization 1-Year Follow-Up Study
Status: Completed | Type: Observational
Sponsor: CryoLife, Inc. (Industry)
Responsible Party: Sponsor
Organization: CryoLife (Unknown)
Other Study IDs: TMR1501.001-M (10/15)
Record Dates: First submitted 2016-02-22; First posted 2016-03-01 (Estimated); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Class IV Angina
Keywords: Angina Pectoris; Angina, Stable; Chest Pain
MeSH Terms: conditions — Angina Pectoris; Angina, Stable; Chest Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Registry Group: Patients previously enrolled in the ANGINA RELIEF Registry who are eligible for a 1-year, prospective follow-up (date of ANGINA RELIEF Registry TMR procedure performed within 12-18 month follow-up window).
- Prospective Group: A group of up to 100 new, prospectively enrolled patients from active centers that receive TMR with the CardioGenesis Laser System and complete a 30-day and 1-year follow-up.

SUMMARY:
The purpose of this study it to collect real world 30-day and 1-year follow-up data for patients undergoing TMR with the CardioGenesis Holmium:YAG Laser System either as a sole therapy procedure or in conjunction with coronary artery bypass graft (CABG) surgery.

The primary objective of this study is to provide ongoing clinical data regarding the characteristics of the patient population undergoing TMR in community practices. Secondary objectives include rates of postoperative mortality and MACE at 30-days and 1-year, and benefit of sustained improvement in angina at 30-days and 1-year.

The study includes two patient populations:

* Registry Group: Patients from selected centers who previously participated in the ANGINA RELIEF Registry and are eligible for a one-year, prospective follow-up;
* Prospective Group: Up to 100 new, prospectively enrolled TMR patients from selected centers.

DETAILED DESCRIPTION:
The study objectives are as follows:

* Track "real world" performance outcomes and physician experience using the CardioGenesis Laser System;
* Further define the disease characteristics of the population being treated;
* Examine transmyocardial revascularization (TMR) usage characteristics, including surgical procedure information, and 30-day and 1-year outcomes;
* Further assess the risk factors for adverse events at 30-days and 1-year;
* Further define MACE rates and angina scores at 30-days and 1-year. To limit the potential for bias, all patients eligible for TMR treatment who meet the Inclusion and Exclusion Criteria will be offered the opportunity to enroll in the study at participating centers.

Primary Endpoint:

- 1-year Canadian Cardiovascular Society (CCS) angina class

Secondary Endpoints:

* All-cause mortality at 30-day and 1-year.
* Rates of major adverse cardiovascular events (MACE) at 30-days and 1-year, defined as the incidence of cardiac-related death, myocardial infarction (Q-wave and non Q-wave), congestive heart failure, cerebrovascular accident, and serious arrhythmia.

The definitions for MACE events are as follows:

* Cardiac-related death: any death that is not clearly attributable to a non-cardiac cause, and includes death due to any of the following: acute myocardial infarction, heart failure, cardiogenic shock, pulmonary edema, cardiac tamponade, arrhythmia, or post-procedural complications (i.e., bleeding).
* Q-wave myocardial infarction: the appearance of new Q waves of 40 or more milliseconds in 2 or more contiguous leads and elevation of CK-MB.
* Non Q-wave myocardial infarction: the elevation of total CK more than twice normal with elevated CK-MB.
* Congestive heart failure: Symptoms of pulmonary vascular congestion or a low output state that is due to left ventricular failure and is new in onset or results in re-hospitalization.
* Cerebrovascular accident: Any sudden development of neurological deficits due to vascular lesions of the brain such as hemorrhage, embolism, or thrombosis that persists for > 24 hours.
* Serious arrhythmia: Supra-ventricular or ventricular arrhythmias that require sustained intravenous pharmacologic treatment, temporary or permanent pacing, or immediate electrical cardioversion or defibrillation. Arrhythmias resulting in syncope, myocardial ischemia, or death are also classified as serious.
* Any other serious operative complications related to the procedure: example: major bleeding requiring transfusion.

ELIGIBILITY:
Inclusion Criteria:

* Registry Group: Previously enrolled in the ANGINA RELIEF Registry; Eligible for a 1-year prospective follow-up (date of TMR procedure performed within 12-18 month follow-up window).
* Prospective Group: Received TMR with the CardioGenesis Laser System; Class IV angina (according to Canadian Cardiovascular Society Angina Scale) prior to TMR; Patients with regions of myocardium in the distal two-thirds of the left ventricle with reversible ischemia and who are not eligible for direct coronary revascularization (e.g., CABG or PTCA).

Exclusion Criteria:

* Registry Group: Date of ANGINA RELIEF Registry TMR procedure performed outside 1-year (12-18 month) follow-up window.
* Prospective Group: Age less than 18 years; Severely unstable angina (un-weanable from intravenous anti-anginals for 48-hours).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who meet the eligibility criteria at the selected centers will be provided an opportunity to participate.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Change in Canadian Cardiovascular Society (CCS) Angina Class from Baseline (Class IV) at 1 Year. | 1 year
  Class I: Ordinary physical activity does not cause angina, such as walking and climbing stairs. Angina with strenuous or rapid or prolonged exertion at work or recreation; Class II: Slight limitation of ordinary activity. Walking or climbing stairs rapidly, walking uphill, walking or stair climbing after meals, or in cold, or in wind, or under emotional stress, or only during the few hours after awakening. Walking more than two blocks on the level and climbing more than one flight of ordinary stairs at a normal pace and in normal conditions; Class III: Marked limitation of ordinary physical activity. Walking one or two blocks on the level and climbing one flight of stairs in normal conditions and at normal pace; Class IV: Inability to carry on any physical activity without discomfort, anginal syndrome may be present at rest.

SECONDARY OUTCOMES:
Rate of all cause mortality | 30 days, 1 year
  All-cause mortality
Rates of Major Adverse Cardiovascular Events (MACE) | 30 days, 1 year
  Defined as the incidence of cardiac-related death, myocardial infarction (Q-wave and non Q-wave), congestive heart failure, cerebrovascular accident, and serious arrhythmia.

CONTACTS AND LOCATIONS:
Overall Officials: Scott B Capps, MS, Study Director — CryoLife, Inc.
Locations (2):
- United States (2):
  - Cardiothoracic and Vascular Surgical Associates, Jacksonville, Florida
  - TriStar Cardiovascular Surgery, Nashville, Tennessee